CLINICAL TRIAL: NCT02942888
Title: The Effects of NAD on Brain Function and Cognition
Brief Title: The Effects of Nicotinamide Adenine Dinucleotide (NAD) on Brain Function and Cognition
Acronym: NAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: University of Texas (Other); South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: HSC20160350H
Record Dates: First submitted 2016-08-29; First posted 2016-10-24 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Mild Cognitive Impairment; NAD
Keywords: Mild Cognitive Impairment; MCI; NAD; nicotinamide riboside; aging
MeSH Terms: conditions — Cognitive Dysfunction | interventions — nicotinamide-beta-riboside; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy control (Active Comparator): Oral administration of NAD precursor, nicotinamide riboside (Niagen; Chromadex Inc.) Dosing will consist of 250mg (week 1), 500mg (week 2), 750mg (week 3), 1g (weeks 4-10). Controls will receive sugar pills.
  Interventions: Dietary Supplement: Nicotinamide riboside; Dietary Supplement: Sugar Pill
- MCI (Experimental): Oral administration of NAD precursor, nicotinamide riboside (Niagen; Chromadex Inc.) Dosing will consist of 250mg (week 1), 500mg (week 2), 750mg (week 3), 1g (weeks 4-10).Controls will receive sugar pills.
  Interventions: Dietary Supplement: Nicotinamide riboside; Dietary Supplement: Sugar Pill

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside — Oral administration of Niagen ramp up 250mg to 1g/day as tolerated
  Other Names: Niagen; ChromaDex, Inc.
Dietary Supplement: Sugar Pill — This is a placebo compounded by ChromaDex, Inc.

SUMMARY:
The purpose of this study is to determine the effects of Niagen (nicotinamide riboside, vitamin B3), on NAD levels, brain function including cognition and blood flow in people diagnosed with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
Niagen is a patented formula which is the first and only commercially available form of Nicotinamide Riboside (NR). It has been proven in basic science studies as a highly effective NAD booster, but it also works as a vitamin B3 supplement. NAD helps pass energy from glucose to other pathways in the cell. Niagen (Nicotinamide Riboside, vitamin B3) is one of the most effective NAD+ precursors to support cellular health.

The purpose of this study is to determine the effects of Niagen (nicotinamide riboside, vitamin B3), on NAD levels, brain function including cognition and blood flow in people diagnosed with mild cognitive impairment (MCI).

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with MCI based on inclusion criteria of Texas Alzheimer's Research Care and Consortium (TARCC) study (IRB: HSC20090535H). We are enrolling both genders, all races and ethnic groups.
* Two week washout period for participants who were taking opioids or a dose of niacin over 200mg

Exclusion Criteria:

* Previously considered as healthy individuals without a MCI or Alzheimer's disease diagnosis based on exclusion criteria of the TARCC study (IRB: HSC20090535H).
* Neurological, psychiatric or active systemic medical disease
* Diabetes
* Moderate or severe depression and/or anxiety as determined the Geriatric Depression Scale (GDS) and the Geriatric Anxiety Scale (GAS), respectively
* Diagnosis of dementia
* Hearing, vision, motor or language deficits
* Alcohol or drug abuse
* Implantation of metal devices
* Administration of Alzheimer's drugs, anticholinergics, neuroleptics, anticonvulsants, opiates, systemic steroids, and mood-stabilizers.
* No opioid use while participating in study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Assessment - Montreal Cognitive Assessment (MoCA) - from baseline at 10 weeks | 10 weeks
  MoCA Value

SECONDARY OUTCOMES:
Change in cerebral blood flow from baseline at 10 weeks | 10 weeks
  functional Magnetic Resonance Imaging (fMRI)
Change in plasma NAD from baseline at 10 weeks | 10 weeks
  Plasma NAD level
Change in Physical Performance - Short Physical Performance Battery (SPPB) - from baseline at 10 weeks | 10 weeks
  SPPB Score
Change in Physical Performance - Instrumental Activities of Daily Living (IADLs) - from baseline at 10 weeks | 10 weeks
  IADL Score
Change in endothelial function from baseline at 10 weeks | 10 weeks
  Arterial Pressure
Change in Cognitive Assessment - Geriatric Depression Scale (GDS) - from baseline at 10 weeks | 10 weeks
  GDS Value (>/= 5 is abnormal)
Change in Cognitive Assessment - Geriatric Anxiety Scale (GAS) - from baseline at 10 weeks | 10 weeks
  GAS Value (Raw score 1 -30)
Change in Cognitive Assessment - Clock Drawing Task Protocol (CLOX) - from baseline at 10 weeks | 10 weeks
  CLOX Value (Score 0-15)
Change in Cognitive Assessment - Executive Interview (EXIT) - from baseline at 10 weeks | 10 weeks
  EXIT Value (Score 0-50)
Change in Cognitive Assessment - Test of Auditory Processing Skills (TAPS) - from baseline at 10 weeks | 10 weeks
  TAPS Score
Change in Physical Performance - Grip Strength - from baseline at 10 weeks | 10 weeks
  Grip Strength (kgs)

CONTACTS AND LOCATIONS:
Overall Officials: Becky Powers, M.D., Principal Investigator — University of Texas Health Science Center in San Antonio
Locations (2):
- United States (2):
  - South Texas Veterans Healthcare System (STVHCS), San Antonio, Texas
  - University of Texas Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orr ME, Kotkowski E, Ramirez P, Bair-Kelps D, Liu Q, Brenner C, Schmidt MS, Fox PT, Larbi A, Tan C, Wong G, Gelfond J, Frost B, Espinoza S, Musi N, Powers B. A randomized placebo-controlled trial of nicotinamide riboside in older adults with mild cognitive impairment. Geroscience. 2024 Feb;46(1):665-682. doi: 10.1007/s11357-023-00999-9. Epub 2023 Nov 23. PMID 37994989